CLINICAL TRIAL: NCT02669563
Title: An Exploratory Study of 18F-Labeled Hydroxyphenethylguanidines in Heart Failure Patients
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, David M. Raffel, Ph.D., Research Associate Professor, University of Michigan
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HUM00105110
Record Dates: First submitted 2016-01-22; First posted 2016-02-01 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathies | interventions — 4-fluoro-3-hydroxyphenethylguanidine; 3-hydroxyephedrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (2):
- Stage 1 (Experimental): Subjects (n = 4 to 10) will be injected once with 20 mCi of [13N]ammonia and receive a 20 minute PET scan. They will then be injected once with 6.5 mCi of one of the two new drugs under study, [18F]4F-MHPG or [18F]3F-PHPG, and receive a 60 minute PET scan.
  On a second visit to the clinic, subjects will be injected once with 6.5 mCi of [18F]3F-PHPG or [18F]4F-MHPG (whichever was not used for the first visit) and receive a 60 minute PET scan.
  Interventions: Drug: [18F]4F-MHPG; Drug: [18F]3F-PHPG; Drug: [13N]ammonia
- Stage 2 (Experimental): Subjects (n = 20 to 26) will be injected with 20 mCi of [13N]ammonia and receive a 20 minute PET scan.
  They will then be injected once with 6.5 mCi of [18F]4F-MHPG or [18F]3F-PHPG (whichever was chosen based on Stage 1 of the study) and receive a 60 minute PET scan. On a second visit to the clinic, subjects will be injected once with 20 mCi of [11C]HED and receive a 40 minute scan.
  Interventions: Drug: [18F]4F-MHPG; Drug: [18F]3F-PHPG; Drug: [13N]ammonia; Drug: [11C]HED

INTERVENTIONS:
Drug: [18F]4F-MHPG — IV injection of [18F]4F-MHPG
  Other Names: 4-[18F]fluoro-meta-hydroxyphenethylguanidine
Drug: [18F]3F-PHPG — IV injection of [18F]3F-PHPG
  Other Names: 3-[18F]fluoro-para-hydroxyphenethylguanidine
Drug: [13N]ammonia — IV injection of [13N]ammonia
  Other Names: [13N]NH3
Drug: [11C]HED — IV injection of [11C]HED
  Other Names: [11C]meta-hydroxyephedrine
  Arms: Stage 2

SUMMARY:
The main goal of this study is to test two new radioactive drugs, 4-[18F]fluoro-meta-hydroxyphenethylguanidine ([18F]4F-MHPG) and 3-[18F]fluoro-para-hydroxyphenethylguanidine ([18F]3F-PHPG) in human subjects with congestive heart failure.

Evaluations of these imaging agents will include their uptake in heart, lungs and liver, their metabolic breakdown in blood, and their kinetics in the heart. Based on these studies, the better of the two drugs will be chosen for further studies in patients with heart disease. After the better compound is chosen, additional measures of its imaging properties, metabolism and pharmacokinetics will be done in subjects with heart failure.

DETAILED DESCRIPTION:
The human heart contains many nerve fibers that are involved in controlling the heart's pumping function. Several heart diseases have been shown to damage the nerves in the heart. Studies have shown that damage to the heart nerves may be a cause of death in patients with diseases like heart failure or diabetes.

Two new radioactive drugs been developed at the University of Michigan for taking pictures of the nerve fibers in the heart using a medical imaging method called positron emission tomography (PET).

These two drugs are 4-[18F]fluoro-meta-hydroxyphenethylguanidine ([18F]4F-MHPG) and 3-[18F]fluoro-para-hydroxyphenethylguanidine ([18F]3F-PHPG). Initial PET imaging studies in normal human subjects (see NCT 02385877) have shown that [18F]4F-MHPG and [18F]3F-PHPG are each able to provide a detailed regional map of the distribution of nerve fibers in the heart.

In Stage 1 of this study, enrolled subjects with heart failure will undergo PET studies with [18F]4F-MHPG and [18F]3F-PHPG to allow direct comparison of the imaging properties, metabolism and pharmacokinetics of the two radioactive drugs in the same subjects.

A third PET scan with [13N]ammonia will be done to assess resting blood flow in different areas of the heart. The results of these studies will be used to select the better of the two tracers for further study in patients with heart disease.

In Stage 2 of the study, enrolled subjects with heart failure will undergo additional PET evaluations of the imaging properties and kinetics of the cardiac nerve tracer selected in Stage 1 (either [18F]4F-MHPG or [18F]3F-PHPG).

Again, a PET scan with [13N]ammonia will also be performed to measure regional resting blood flow. A third PET scan with [11C]meta-hydroxyephedrine ([11C]HED), an established cardiac nerve tracer, will also be done to address research questions related to the mechanisms involved in the retention of [18F]4F-MHPG and [18F]3F-PHPG inside the nerve of the heart.

For all study stages, subjects will be assessed during the scan for heart rate, blood pressure and oxygen saturation. Patients will be followed at 30 min, 24 hours and 30 hours regarding any adverse events or serious adverse events they might have experienced. These will be reported as required.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80y
* Cardiomyopathy (ischemic and non-ischemic)
* Left ventricular ejection fraction (LVEF) < 35%
* Clinically appropriate referral for surgical implantation of an implantable cardiodefibrillator (ICD) for primary prevention of sudden cardiac death
* Not claustrophobic
* Ability to lie flat for 90 min
* Give informed consent

Exclusion Criteria:

* Revascularization such as the placement of a stent or balloon angioplast in the preceding 40 days
* Renal dysfunction with eGFR < 50 mL/min/1.73 m2
* Currently taking medications or drugs that may alter PET scans of cardiac sympathetic nerve terminals with these tracers, including any of the following:

  * Tricyclic antidepressants, which inhibit the norepinephrine transporter, such as amitriptyline, desipramine, imipramine, etc.
  * Cold medications (e.g., Sudafed®, as they may contain sympathomimetic amines, such as phenylephrine, phenylpropanolamine, pseudoephedrine, etc.)
  * Nasal decongestants (some use phenylephrine as the active agent)
  * Cocaine (which inhibits the norepinephrine transporter)
  * Tetrabenazine (Xenazine, which inhibits VMAT2 transporters on vesicles inside neurons)
  * Monoamine oxidase inhibitors (MAOI)
  * Some antihypertensive drugs (reserpine, labetalol, α-methyldopa, and clonidine)
* Pregnancy or lactation
* Claustrophobia
* Inability to lie flat for 90 min

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-12; Primary Completion 2016-08 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Composite measures based on radiotracer tissue uptake ratios (heart-to-lung ratio, heart-to-liver ratio, heart-to-blood ratio) and rates of metabolism in plasma (half-time, minutes) of [18F]4F-MHPG and [18F]3F-PHPG in patients with heart failure. | 12 months
  These data on the relative imaging properties and metabolism of [18F]4F-MHPG and [18F]3F-PHPG in heart failure patients will be used to select the lead radiotracer for further clinical development.

SECONDARY OUTCOMES:
Quantitative measures of regional cardiac sympathetic nerve density in patients with heart failure using tracer kinetic analyses. | 36 months
  Robust metrics of regional sympathetic nerve density in the heart obtained using tracer kinetic analysis techniques, including compartmental modeling and Patlak graphical analysis, will contribute to selection of a lead radiotracer.
Number of study participants with adverse events as a measure of safety and tolerability following intravenous administration of [18F]4F-MHPG or [18F]3F-PHPG. | Up to 30 days after [18F]4F-MHPG or [18F]3F-PHPG injection.
  Assessments of the safety of [18F]4F-MHPG and [18F]3F-PHPG as PET radiopharmaceuticals for routine studies in patients.

CONTACTS AND LOCATIONS:
Overall Officials: David M Raffel, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Raffel DM, Crawford TC, Jung YW, Koeppe RA, Gu G, Rothley J, Frey KA. Quantifying cardiac sympathetic denervation: first studies of 18F-fluorohydroxyphenethylguanidines in cardiomyopathy patients. Eur J Nucl Med Mol Imaging. 2022 Jan;49(2):619-631. doi: 10.1007/s00259-021-05517-7. Epub 2021 Aug 13. PMID 34387718